CLINICAL TRIAL: NCT04612751
Title: A Phase 1b, Multicenter, 2-Part, Open-Label Study of Datopotamab Deruxtecan (Dato-DXd) in Combination With Immunotherapy With or Without Carboplatin in Participants With Advanced or Metastatic Non-Small Cell Lung Cancer (Tropion-Lung04)
Brief Title: Phase 1b Study of Dato-DXd in Combination With Immunotherapy With or Without Carboplatin in Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: TROPION-Lung04
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D926FC00001; 2023-505992-54-00 (Registry Identifier: CTIS (EU)); 2021-000274-28 (EudraCT Number)
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic NSCLC
Keywords: Advanced or Metastatic NSCLC; Datopotamab deruxtecan (Dato-DXd); DS-1062a; Durvalumab; AZD2936; MEDI5752; AZD7789
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Cohort 1 (Experimental): Datopotamab deruxtecan (Dato-DXd) + Durvalumab in NSCLC participants who are either treatment-naïve or have received only 1 prior line of systemic chemotherapy without concomitant ICI therapy
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab
- Cohort 2 (Experimental): Datopotamab deruxtecan (Dato-DXd) + Durvalumab in NSCLC participants who are either treatment-naïve or have received only 1 prior line of systemic chemotherapy without concomitant ICI therapy
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab
- Cohort 3 (Experimental): Datopotamab deruxtecan (Dato-DXd) + Durvalumab + Carboplatin in NSCLC participants who are either treatment-naïve or have received only 1 prior line of systemic chemotherapy without concomitant ICI therapy
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab; Drug: Carboplatin
- Cohort 4 (Experimental): Datopotamab deruxtecan (Dato-DXd) + Durvalumab + Carboplatin in NSCLC participants who are either treatment-naïve or have received only 1 prior line of systemic chemotherapy without concomitant ICI therapy
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab; Drug: Carboplatin
- Cohort 5 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD2936 in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: AZD2936
- Cohort 6 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD2936 in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: AZD2936
- Cohort 7 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD2936 + Carboplatin in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: Carboplatin; Drug: AZD2936
- Cohort 8 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD2936 + Carboplatin in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: Carboplatin; Drug: AZD2936
- Cohort 9 (Experimental): Datopotamab deruxtecan (Dato-DXd) + MEDI5752 + Carboplatin in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: Carboplatin; Drug: MEDI5752
- Cohort 10 (Experimental): Datopotamab deruxtecan (Dato-DXd) + MEDI5752 + Carboplatin in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: Carboplatin; Drug: MEDI5752
- Cohort 11 (Experimental): Datopotamab deruxtecan (Dato-DXd) + MEDI5752 in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: MEDI5752
- Cohort 12 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD7789 in participants with CPI acquired resistant NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: AZD7789
- Cohort 13 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD7789 in participants with CPI acquired resistant NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: AZD7789
- Cohort 14 (Experimental): Datopotamab deruxtecan (Dato-DXd) + AZD7789 in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: AZD7789
- Cohort 4A (Experimental): Datopotamab deruxtecan (Dato-DXd) + Durvalumab + carboplatin in participants with treatment-naïve NSCLC
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Datopotamab deruxtecan — Intravenous infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle
  Other Names: Dato-DXd
Drug: Durvalumab — Intravenous infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle
  Other Names: Imfinzi
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 4A
Drug: Carboplatin — Intravenous infusion Q3W on Day 1 or Day 2 of each 21-day cycle
  Arms: Cohort 10; Cohort 3; Cohort 4; Cohort 4A; Cohort 7; Cohort 8; Cohort 9
Drug: AZD2936 — Intravenous infusion prior to Dato-DXd every 3 weeks (Q3W) on Day 1 prior to Dato-Dxd of each 21-day cycle
  Other Names: rilvegostomig
  Arms: Cohort 5; Cohort 6; Cohort 7; Cohort 8
Drug: MEDI5752 — Intravenous infusion prior to Dato-DXd every 3 weeks (Q3W) on Day 1 prior to Dato-Dxd of each 21-day cycle
  Other Names: volrustomig
  Arms: Cohort 10; Cohort 11; Cohort 9
Drug: AZD7789 — Intravenous infusion prior to Dato-DXd every 3 weeks (Q3W) on Day 1 prior to Dato-Dxd of each 21-day cycle
  Other Names: sabestomig
  Arms: Cohort 12; Cohort 13; Cohort 14

SUMMARY:
This study will assess safety, tolerability, and treatment activity of datopotamab deruxtecan (Dato-DXd) in combination with immunotherapy with or without carboplatin in participants with advanced or metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The primary objective is to assess the safety and tolerability of Dato-DXd in combination with immunotherapy with or without 4 cycles of carboplatin in participants with advanced or metastatic NSCLC.

Two dose levels of Dato-DXd will be studied in combination with immunotherapy (durvalumab, AZD2936, MEDI5752, or AZD7789) with or without 4 cycles of carboplatin in 15 study cohorts

Each cohort will start with Part 1 (dose escalation or confirmation), where 3 to 9 participants will be assessed for dose-limiting toxicities (DLT) in the first cycle of treatment. if the DLT incidence rate meets the criteria based on the modified toxicity probability interval-2 (mTPI-2), then Part 2 (dose expansion) may be opened.

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥18 years old on the day of signing the ICF (local regulatory requirement to consent should be followed).
* Histologically or cytologically confirmed diagnosis of advanced or metastatic NSCLC, without EGFR or ALK genomic alterations (testing not required for participants with documented squamous histology) and no known genomic alterations in other actionable driver kinases with approved therapies. Participants whose tumors harbor KRAS mutations are eligible for this study.
* For Cohorts 1 to 4, participants must be treatment-naïve or have received and radiologically progressed after only 1 prior line of systemic chemotherapy, without concomitant immune checkpoint inhibitors for advanced or metastatic NSCLC. For Cohorts 4a, 5 to 11, and 14, participants must be treatment-naïve for advanced or metastatic NSCLC. For Cohorts 12 to 13, participants must be CPI acquired resistant after 1 or 2 prior lines of systemic therapy for advanced or metastatic NSCLC, of which 1 should have contained an approved anti-PD-1/PD L1. Cohort 4a will enroll participants whose tumors have squamous histology only; Cohorts 5 Part 2A and Part 2B as well as Cohorts 12 and 13 will enroll participants whose tumors have non-squamous histology only.
* Willing and able to undergo a mandatory tumor biopsy. A tumor biopsy that was recently collected (within 3 months of screening) after completion of the most recent anticancer treatment regimen may be substituted for the biopsy collected during screening. For Cohorts 12 and 13, a tumor sample taken ≤24 months prior to screening is acceptable.
* Has measurable disease per RECIST1.1 within 28 days prior to Cycle 1 Day 1
* Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Has adequate bone marrow reserve and organ function at baseline within 7 days prior to Cycle 1 day 1
* For Cohorts 5 to 14 only: Documented IHC PD-L1 expression per analytically validated Ventana PD-L1 (SP263) IHC assay, 22C3 PharmDx assay, or 28-8 PharmDx assay

Exclusion Criteria:

* Active or prior documented autoimmune or inflammatory disorders
* Uncontrolled or significant cardiac disease
* History of another primary malignancy with exceptions
* active or uncontrolled hepatitis B or C virus or uncontrolled HIV infection
* spinal cord compression or clinically active CNS metastases
* History of (non-infectious) ILD/pneumonitis that required steroids
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illness
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Clinically significant corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with DLTs; TEAEs and other safety parameters during the study. | DLTs: within first cycle (21 days); TEAEs and other safety parameters: when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up (approximately 60 months)
  DLTs, TEAEs, SAEs, AESIs, ECOG PS, vital sign measurements, standard clinical laboratory parameters (hematology, clinical chemistry, and urinalysis), ECG parameters, ECHO/MUGA scan findings, and ophthalmologic findings

SECONDARY OUTCOMES:
ORR as assessed by investigator per RECIST Version 1.1 | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  ORR is defined as the proportion of participants with measurable disease at baseline who achieved a BOR of confirmed CR or confirmed PR.
Duration of Response as assessed by investigator per RECIST version 1.1 | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Duration of Response is defined as the time from the date of the first documentation of objective response (confirmed CR or confirmed PR) to the date of the first documentation of objective PD, or death due to any cause, whichever occurs first.
Disease Control Rate as assessed by the investigator per RECIST version 1.1 | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Disease Control Rate is defined as the proportion of participants who achieved a Best Overall Response of confirmed complete response, confirmed partial response, or stable disease.
Progression-free Survival as assessed by the investigator per RECIST v1.1 | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Progression-free Survival is defined as the time interval from the date of the start of study treatment to the earlier of the dates of the first documentation of objective PD or death due to any cause, whichever occurs first
Time to Response as assessed by investigator per RECIST Version 1.1 | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Time to Response is defined as the time from the date of the start of study treatment to the date of the first documentation of objective response (confirmed complete response or confirmed partial response)
Best percentage change in the Sum of Diameters of measurable tumors | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  The best percentage change in the Sum of Diameters of measurable tumors is defined as the percentage change in the smallest Sum of Diameters from all postbaseline tumor assessments, taking as reference the baseline Sum of Diameters.
Overall Survival | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Overall Survival is defined as the time from the date of the start of study treatment to the date of death due to any cause
Pharmacokinetic Parameter Maximum Plasma/Serum Concentration (Cmax) of Dato-DXd, Total anti-TROP2 antibody, and MAAA-1181a. Serum concentrations of durvalumab and MEDI5752, AZD2936, MEDI5752 and AZD7789. | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Cmax = Maximum concentration
Pharmacokinetic Parameter Time to Maximum Plasma/Serum Concentration (Tmax) of Dato-DXd, Total anti-TROP2 antibody, and MAAA-1181a. | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Tmax = time to reach maximum concentration.
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve (AUC) of Dato-DXd, Total anti-TROP2 antibody, and MAAA-1181a. | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  Area under the plasma concentration-time curve up to last quantifiable time (AUClast) and area under the plasma concentration-time curve during dosing interval (AUCtau) will be assessed.
Prevalence of Dato-Dxd, durvalumab, AZD2936, MEDI5752 and AZD7789 ADA | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  ADA prevalence is defined as the proportion of all participants having ADA at any point in time (including pre-existing ADA at baseline and treatment-emergent ADA)
Incidence of Dato-DXd, durvalumab, AZD2936, MEDI5752 and AZD7789 ADA | At the time of the final analysis (when all participants have either discontinued the study or the last participant enrolled in the study has completed at least 9 months of follow-up, approximately 60 months).
  ADA incidence is defined as the proportion of participants having treatment-emergent ADA during the study period

CONTACTS AND LOCATIONS:
Locations (37):
- United States (10):
  - Research Site, La Jolla, California
  - Research Site, Santa Ana, California
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Belgium (2):
  - Research Site, Hasselt
  - Research Site, Roeselare
- Italy (4):
  - Research Site, Aviano
  - Research Site, Meldola
  - Research Site, Orbassano
  - Research Site, Roma
- Japan (3):
  - Research Site, Kōtoku
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Hsinchu
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/257839